CLINICAL TRIAL: NCT03093285
Title: OBSERVATIONAL STUDY FOR EVALUATIING THE EFFECT OF RESTORING Euthyroidism ON FEMALE SEXUAL FUNCTION
Brief Title: Dysthyroidism and Female Sexual Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Mario Maggi, PROFESSOR, University of Florence
Other Study IDs: Andro AOUC 2016 01
Record Dates: First submitted 2017-02-16; First posted 2017-03-28 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Sexuality; Thyroid
MeSH Terms: conditions — Sexuality; Thyroid Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- dysthyoidic female: sexually active, hypothyroidic or hyperthyroidic women of childbearing age

SUMMARY:
The aim of the study is to evaluate the incidence of sexual dysfunction in presence of dysthyroidism and the impact of restoring euthyroidism on female sexual function

DETAILED DESCRIPTION:
Hormonal component plays a crucial role in sexual function. Hypothyroidism and hyperthyroidism may be associated with any form of sexual dysfunction in men but only a few studies reported the relationship between thyroid dysfunction and female sexuality.

The study is an observational study. An informed consent will be obtained from all patients before the study.

The aim of the study is:

* to evaluate the incidence of sexual dysfunction in presence of dysthyroidism and the impact of restoring euthyroidism on female sexual function (evaluated with the Female Sexual Function Index)
* to evaluate the influence of hormonal changes on the emotional and psychological wellness (evalueted with the Middle Sex Hospital Questionnaire)
* to evaluate the influence of hormonal changes on the satisfaction of body image (evalueted with the Body Uneasiness Test)
* to evaluate the influence of hormonal changes on the distress related to sexuality (evaluated with the Female Sexual Distress Scale).

The investigators espect to enroll a total of 50 sexually active hyperthyroidic/hypothyroidic women in this study in about 7 months. Statistical analyses will be performed using the Statistical Package for the Social Sciences

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* hyperthyroidic or hypothyroiditic women
* sexually active women

Exclusion Criteria:

* age < 18 Y
* no sexual activity
* pregnancy
* psychiatric disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: sexually active, hyperthyroidic or hypothyroiditic women
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Sexual Dysfunction and dysthyroidism | 12 months
  To assess the incidence of sexual dysfunction in the presence of dysthyroidism and the impact of restoring euthyroidism on female sexual function. The investigators will evaluate the difference between the scores of the FSFI (Female Sexual Function Index) questionnaire administered at baseline and after normalization of thyroid function. The test consists of six domains: desire, arousal, orgasm, pain, sexual satisfaction, lubrication. For each domain the total score goes from 0 to 6 (full sexual functionality).

SECONDARY OUTCOMES:
Weelbeing and dysthyroidism | 12 months
  To evaluate the influence of hormonal changes on the emotional and psychological wellbeing considering the difference between the scores of the MHQ (Middle Sex Hospital Questionnaire) questionnaire administered at baseline and after normalization of thyroid function. The MHQ test is a self-administered questionnaire used for screening of mental disorders. It consists of six areas related to the free anxiety, phobic anxiety, obsessive compulsive symptoms, somatization, depressive symptoms and histrionic-hysterical traits.
Body image and dysthyroidism | 12 months
  To evaluate the influence of hormonal changes on the satisfaction of body image considering the difference between the scores of the BUT (Body Uneasiness Test) questionnaire administered at baseline and after normalization of thyroid function. The test consists of two parts (A and B) which respectively evaluate the degree of severity linked to body image and some sensory events derived from a precise area of the body. A reduction of the score between the baseline and the normalization of thyroid function would indicate an improvement in these aspects.
Distress related to sexuality and dysthyroidism | 12 months
  To evaluate the influence of hormonal changes on the distress related to sexuality considering the difference between the scores of the FSDS (Female Sexual Distress Scale Revised) questionnaire administered at baseline and after normalization of thyroid function. A higher score (0-48) represents a greater sexual distress.

CONTACTS AND LOCATIONS:
Overall Officials: mario maggi, MD, Study Director — Andrology Unit
Locations (1):
- Andrology Unit, Florence, Italy

REFERENCES:
- [Result] Atis G, Dalkilinc A, Altuntas Y, Atis A, Caskurlu T, Ergenekon E. Sexual dysfunction in women with clinical hypothyroidism and subclinical hypothyroidism. J Sex Med. 2010 Jul;7(7):2583-90. doi: 10.1111/j.1743-6109.2010.01815.x. Epub 2010 Apr 20. PMID 20412428
- [Result] Battaglia C, Nappi RE, Mancini F, Cianciosi A, Persico N, Busacchi P, Facchinetti F, de Aloysio D. Menstrual cycle-related morphometric and vascular modifications of the clitoris. J Sex Med. 2008 Dec;5(12):2853-61. doi: 10.1111/j.1743-6109.2008.00972.x. Epub 2008 Aug 28. PMID 18761595
- [Result] Bhasin S, Enzlin P, Coviello A, Basson R. Sexual dysfunction in men and women with endocrine disorders. Lancet. 2007 Feb 17;369(9561):597-611. doi: 10.1016/S0140-6736(07)60280-3. PMID 17307107
- [Result] Crown S, Crisp AH. A short clinical diagnostic self-rating scale for psychoneurotic patients. The Middlesex Hospital Questionnaire (M.H.Q.). Br J Psychiatry. 1966 Sep;112(490):917-23. doi: 10.1192/bjp.112.490.917. No abstract available. PMID 5970912
- [Result] Derogatis L, Clayton A, Lewis-D'Agostino D, Wunderlich G, Fu Y. Validation of the female sexual distress scale-revised for assessing distress in women with hypoactive sexual desire disorder. J Sex Med. 2008 Feb;5(2):357-64. doi: 10.1111/j.1743-6109.2007.00672.x. Epub 2007 Nov 27. PMID 18042215
- [Result] Krassas GE. Thyroid disease and female reproduction. Fertil Steril. 2000 Dec;74(6):1063-70. doi: 10.1016/s0015-0282(00)01589-2. PMID 11119728
- [Result] Oppo A, Franceschi E, Atzeni F, Taberlet A, Mariotti S. Effects of hyperthyroidism, hypothyroidism, and thyroid autoimmunity on female sexual function. J Endocrinol Invest. 2011 Jun;34(6):449-53. doi: 10.1007/BF03346712. Epub 2011 Apr 28. PMID 21532331
- [Result] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451